CLINICAL TRIAL: NCT04459143
Title: Chronic Obstructive Pulmonary Disease (COPD) and Advance Directives
Acronym: DIABPCO
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD 0918
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Palliative care; Advance directives; Exacerbation; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Advance Directives

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Advance directives — A workshop will take place during the third week of patient care to inform them about COPD, exacerbations, prognostic and advance directives. Then, a personal interview with patients who have participated to this workshop will take place at the end of their hospital stay, to collect their advance directives and their degree of satisfaction about this process.

SUMMARY:
The aim of this study is to evaluate if the participation of COPD patients to a workshop on advance directives increases the number of patients who write them.

DETAILED DESCRIPTION:
Chronic Obstructive Disease is a common disease and should be the third leading cause of death in 2020. Patient hospitalized for an exacerbation of their COPD have a median survival of 2 years and 50% risk of being rehospitalized within 6 months.

COPD patients may have symptoms that impair their life quality significantly and sometimes more than patients with cancer. This is particularly the case for dyspnea, which is frequently present.

In the study, Investigators propose the setting up of health workshop on advance directives. This workshop is for sever or very severe COPD patients during their hospital stay in the post-acute care and pulmonary rehabilitation service.

In this unit, investigators welcome patient from all the region of Ile de France for a hospital stay of approximately 6 weeks. A first workshop will take place during the third week of their care to inform them about COPD, exacerbations, prognostic and advance directives. Then, a personal interview with patients who have participated to this workshop will take place to collect their advance directives and their degree of satisfaction about this process.

ELIGIBILITY:
Inclusion Criteria:

* COPD Gold 3 or 4 and Curtis criteria

Exclusion Criteria:

* left to the discretion of the investigator if he finds that it will not be beneficial for the patient : for example if the workshop is judged to be at risk of being anxiety-provoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with COPD Gold 3 or 4 who accept to participate to the workshop
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patient who write their advance directives | At the end of patient hospital stay, approximately 6 weeks
  The Primary Outcome Measure is the collect of the number of patients who write their advance directives after their participation of the health workshop

SECONDARY OUTCOMES:
Measure of patient's satisfaction | At the end of patient hospital stay, approximately 6 weeks
  The satisfaction of patient was measured with a satisfaction questionnaire scale based on their feelings about the workshop. For each item, patient ticks : Strongly agree, Agree, Neither agree or disagree, Disagree or Strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Boitiaux, Principal Investigator — Hôpital NOVO
Locations (1):
- Les Cèdres SSR Pneumologie / Réhabilitation Respiratoire, Aincourt, France